CLINICAL TRIAL: NCT03704402
Title: Effect of High School Alcohol Policies on Students' Binge Drinking- a Natural Experiment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 15/4155
Record Dates: First submitted 2018-08-10; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Policy; Binge Drinking
MeSH Terms: conditions — Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alcohol policy group: High schools that introduced the policy
  Interventions: Other: Alcohol policy
- control group: High schools that did not introduce the policy

INTERVENTIONS:
Other: Alcohol policy — Introduction of new mutual alcohol policy
  Groups: alcohol policy group

SUMMARY:
The aim of the project is to evaluate the effects of the introduction of new mutual alcohol policies in 30 high schools in 2017 on students binge drinking.

DETAILED DESCRIPTION:
In August 2017, 13 high schools in Zealand and all of Funen's 11 high schools and 6 high schools in Ringkøbing introduced new mutual alcohol policy for alcohol on study trips, parties, cafes and other social events.

The background for the introduction of the alcohol policies was the aim of reducing alcohol intake among students and that alcohol should have a less dominant role. By setting the same framework, the alcohol policies aims at promoting community, responsibility and respect.

The aim of the project is to evaluate the effects of the introduction of new mutual alcohol policies on students binge drinking.

The analysis is a natural experiment that compare binge drinking among students at schools after the introduction of the policy with binge drinking among students a schools that did not introduce the policy.

ELIGIBILITY:
Inclusion Criteria:

* High school student

Exclusion Criteria:

-

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consist of high school students participating in the Danish National Youth Study 2014 and the Danish National High School Study 2019
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Binge drinking 4 or more times within the last month | january 2019
  Reduction in the number of students that drink 5 or more drinks on the same occasion 4 or more times within the last month

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Pisinger, Principal Investigator — Southern Denmark University

IPD SHARING:
Plan to Share IPD: No